CLINICAL TRIAL: NCT00061958
Title: A Phase II Study of Arsenic Trioxide (NSC 706363) in Patients With Advanced Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Arsenic Trioxide in Treating Patients With Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02534; DM02-172; N01CM17003 (NIH); CDR0000302483 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Esophagus; Stage III Esophageal Cancer; Stage IV Esophageal Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Arsenic Trioxide

ARMS (1):
- Treatment (arsenic trioxide) (Experimental): Patients receive a loading dose of arsenic trioxide IV over 2 hours on days 1-5 on week 1. Beginning on week 2, patients receive a maintenance dose of arsenic trioxide IV twice weekly thereafter. Courses repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients achieving a CR continue to receive therapy for at least 6 months beyond CR.
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox

SUMMARY:
This phase II trial is studying how well arsenic trioxide works in treating patients with metastatic or unresectable cancer of the esophagus or gastroesophageal junction. Drugs used in chemotherapy such as arsenic trioxide use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate and duration of response in patients with advanced adenocarcinoma of the esophagus or gastroesophageal junction treated with arsenic trioxide.

II. Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive a loading dose of arsenic trioxide IV over 2 hours on days 1-5 on week 1. Beginning on week 2, patients receive a maintenance dose of arsenic trioxide IV twice weekly thereafter. Courses repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) continue to receive therapy for at least 6 months beyond CR.

Patients are followed every 3 months for 6 months or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * Metastatic or unresectable local-regional disease
  * Osseous metastasis as the only site of disease not eligible
* Measurable disease

  * Mediastinal or hilar lymph nodes must be at least 2.0 cm in diameter by CT scan or MRI to be considered measurable
* No known brain metastases
* Performance status - Zubrod 0-2
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL
* Bilirubin no greater than 1.5 mg/dL
* SGOT and/or SGPT no greater than 2.0 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min
* Calcium no greater than 12 mg/dL
* No symptomatic hypercalcemia under treatment
* No New York Heart Association class III or IV heart disease
* No angina within the past 6 months
* No myocardial infarction within the past 6 months
* No congestive heart failure within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Prior malignancies with no evidence of disease for at least 2 years are allowed
* No serious concurrent infection that is uncontrolled or whose control could be jeopardized by complications of study therapy
* No concurrent nonmalignant medical illness that is uncontrolled or whose control could be jeopardized by complications of study therapy
* No psychiatric disorder or other condition that would preclude study compliance
* No prior immunotherapy (including adjuvant or preoperative regimens)
* No concurrent biological response modifiers
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* No prior chemotherapy (including adjuvant or preoperative regimens and radiosensitizers)
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to major bone marrow containing areas (e.g., pelvis or lumbar spine) or area that contained the indicator lesion
* No prior radiotherapy involving 30% or more of the bone marrow
* No concurrent radiotherapy
* At least 2 weeks since prior major surgery (4 days for minor surgery) and recovered
* No other concurrent investigational drugs
* No other concurrent antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-06; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Objective response (OR) defined as a complete or partial remission, evaluated using RECIST criteria | 8 weeks

SECONDARY OUTCOMES:
Duration of response | From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 6 months
Toxicity graded according to the Common Toxicity Criteria version 2 | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States